CLINICAL TRIAL: NCT04696575
Title: A Phase II Trial of Lamivudine in Combination With Chemoimmunotherapy in Patients With Extensive Stage SCLC
Brief Title: Lamivudine in Combination With Chemoimmunotherapy for the Treatment of Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 691720; NCI-2020-13169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 691720 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma
MeSH Terms: interventions — atezolizumab; Carboplatin; Etoposide; Lamivudine; lipoarabinomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (lamivudine, chemoimmunotherapy) (Experimental): INDUCTION: Patients receive lamivudine PO QD on days 1-28. Patients also receive carboplatin IV over 30-60 minutes and atezolizumab IV on day 1, and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive lamivudine PO QD on days 1-28 and atezolizumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  NOTE: Patients who are not eligible for atezolizumab as outlined in exclusion criteria or who refuse to receive atezolizumab may still be treated in this study with carboplatin and etoposide as the IV drug component, in addition to lamivudine orally administered.
  Interventions: Biological: Atezolizumab; Drug: Carboplatin; Drug: Etoposide; Drug: Lamivudine

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Lamivudine — Given PO
  Other Names: (-)-BCH-189; 3TC; Epivir; GR109714X; LAM

SUMMARY:
This phase II trial studies the effect of lamivudine in combination with standard of care chemoimmunotherapy in treating patients with extensive stage small cell lung cancer. Even though small cell lung cancer is initially highly responsive to first-line chemotherapy treatment, treatment resistance inevitably emerges; treatment resistance is when tumor cells stop responding to a drug treatment that they had previously responded to. Lamivudine is an oral antiviral a drug that may be able to reduce the ability of tumors to develop drug resistance. Chemotherapy drugs, such as carboplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving lamivudine together with the usual standard of care chemoimmunotherapy may help prevent the growth and spread of the tumor cells to other parts of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the 6-month progression-free survival (PFS) rate of lamivudine in combination with platinum-based chemotherapy in patients with extensive stage small cell lung cancer (SCLC).

SECONDARY OBJECTIVES:

I. To evaluate the 12-month survival and overall survival (OS) of patients with extensive stage SCLC receiving study treatment.

II. To assess the toxicity of the combination of lamivudine with platinum-based chemotherapy in this population.

EXPLORATORY OBJECTIVE:

I. To study tissue and blood-based biomarkers as potential predictors of treatment outcomes.

OUTLINE:

INDUCTION: Patients receive lamivudine orally (PO) once daily (QD) on days 1-28. Patients also receive carboplatin intravenously (IV) over 30-60 minutes and atezolizumab IV on day 1, and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive lamivudine PO QD on days 1-28 and atezolizumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: Patients who are not eligible for atezolizumab as outlined in exclusion criteria or who refuse to receive atezolizumab may still be treated in this study with carboplatin and etoposide as the IV drug component, in addition to lamivudine orally administered.

After completion of study treatment, patients are followed up for 30 days and then every 60 days thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1 at the time of study treatment initiation
* Histologically or cytologically confirmed diagnosis of small cell lung cancer (SCLC)
* Patient should have extensive stage disease, defined as, malignant pleural effusion, pulmonary metastases in a different lobe in the ipsilateral lung or contralateral lung, and/or the presence of extra-thoracic metastatic disease
* Must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 prior to starting platinum-based systemic chemotherapy
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 x institution upper limit of normal (ULN) and calculated creatinine clearance of at least 15 ml/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN) (ALT and AST =< 5 x ULN is acceptable if liver metastases are present)
* Total serum bilirubin =< 1.5 x ULN. For patients with well documented Gilbert's syndrome, total bilirubin =< 3 x ULN with direct bilirubin within normal range
* Newly diagnosed SCLC patients may receive no more than 1 cycle of standard chemotherapy or chemoimmunotherapy for their current diagnosis prior to study treatment
* Patients who have progressed on prior treatment for SCLC will be eligible if both of the following conditions are met:

  * Received no more than one-line of treatment with platinum-based chemotherapy for SCLC, and
  * Last platinum-based treatment administered >= 12 months prior to diagnosis of recurrence/relapse. Patients should not have experienced disease progression while receiving prior platinum-based treatment for SCLC
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Receipt of anticancer chemotherapy/chemoimmunotherapy within 4 weeks prior to the first administration of study drug other than what is allowed in the inclusion criteria
* Symptomatic brain metastasis

  * Patients with treated brain metastases are eligible provided they have recovered from effects of radiation and neurological symptoms are improved or controlled for at least two weeks prior to enrollment
  * Patients with asymptomatic brain metastases who are being treated with systemic chemotherapy alone are also eligible if no more than 6 lesions each less than 1 cm in size is present at the time of initiating protocol treatment
* Leptomeningeal involvement regardless of treatment status
* Participation in another interventional study within the last 28 days of study enrollment
* Had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered major surgery) resulting from a prior surgery
* Positive for immunosuppressive disease, acquired immunodeficiency syndrome (AIDS) or other immune depressing diseases. For human immunodeficiency virus (HIV), HVC and HBC-mandatory testing is required prior to enrollment

  * Note: Patients with past or resolved hepatitis B virus (HBV) infection (defined as the presence of hepatitis B surface antibody [HBsAb] and absence of hepatitis B surface antigen [HBsAg]) are eligible (HBV deoxyribonucleic acid [DNA] should be obtained in patients if only anti-hepatitis B core [HBc] antibody was present prior to randomization). Patients with active/untreated hepatitis C virus (HCV) will be excluded from the study; patients who test positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Active, clinically serious infections or other serious uncontrolled medical conditions, including chronic viral hepatitis (testing for hepatitis B, C required)
* Patient has known hypersensitivity to the components of the study drugs or any analogs
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

  * Myocardial infarction or arterial or venous thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) class III or IV disease
  * History of documented congestive heart failure (New York Heart Association functional classification III or IV) within 6 months prior to baseline
  * Poorly controlled arrhythmias
* Contraindications to atezolizumab: Patients with active autoimmune disorder or prior history of autoimmune disorder requiring immunosuppressive agents within preceding two years will not be allowed to receive atezolizumab but will be able to receive the other drugs included in the treatment regimen, if eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From the date of registration to the date of first confirmed progression or death, whichever occurred first, assessed at 6 months
  The primary test of efficacy will be carried out using an exact binomial test of a proportion. Descriptive analyses will be carried out using the Kaplan-Meier product-limit estimator. Patients who are treated beyond RECIST progression and subsequently had tumor response while on study (and no other intervening treatment) will be classified as pseudoprogression and not counted as progression event.

SECONDARY OUTCOMES:
Overall survival | From registration to death from any cause or 5 years from time of enrollment, whichever occurs first
  Descriptive analyses will be carried out using the Kaplan-Meier product-limit estimator.
Incidence of toxicities | Up to 30 days after the end of all treatment
  Per National Cancer Institute Common Terminology Criteria for Adverse Events version 5, the term toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded for each patient and will be used for reporting. Frequency tables will be reviewed to determine toxicity patterns. In addition, all adverse event data graded as 3, 4, or 5 and classified as either "unrelated or unlikely to be related" to study treatment in the event of an actual relationship developing will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Grace K Dy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States